CLINICAL TRIAL: NCT04746547
Title: An Open-label, Sequential Non-randomised Pharmacokinetics Study of DTG Plasma Exposure When Given as Twice or Once Daily DTG in the Presence of Rifampicin in Children With HIV and TB Between 20-35kgs in SA
Brief Title: Pharmacokinetics of Twice or Once Daily DTG (50mg) in Children With HIV and TB
Acronym: ORCHID
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of KwaZulu (Other)
Collaborators: Centre for the AIDS Programme of Research in South Africa (Network)
Responsible Party: Principal Investigator, Dr Moherndran Archary, Dr Moherndran Archary, University of KwaZulu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPRISA258 (CAP258)
Record Dates: First submitted 2021-02-01; First posted 2021-02-09 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Tuberculosis; Hiv
Keywords: Dolutegravir (DTG); Paediatrics; HIV/TB co-infection
MeSH Terms: conditions — Tuberculosis; Acquired Immunodeficiency Syndrome | interventions — dolutegravir

STUDY DESIGN:
Intervention Model Description: Pharmacokinetic evaluation of DTG in children receiving Rifampicin containing TB treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Twice Daily DTG (Other): Twice daily Dolutegravir (50mg) with Rifampicin containing TB treatment / Twice daily Dolutegravir (10mg) dispersible
  Interventions: Drug: Dolutegravir 50 MG; Drug: Dolutegravir 10 MG

INTERVENTIONS:
Drug: Dolutegravir 50 MG — Twice daily dolutegravir with rifampicin containing TB treatment
Drug: Dolutegravir 10 MG — Twice daily dolutegravir with rifampicin containing TB treatment

SUMMARY:
Stage 1 proposed study will provide evidence to support the use of twice-daily dose 50mg DTG in children (20-35kgs) co-treated with RIF.

Note: An amendment has been added to include children from 3kgs and a dose of 10mg dispersible DTG

DETAILED DESCRIPTION:
This is a single centre, open-label, non-randomised, prospective study evaluating the steady-state pharmacokinetics of twice-daily dose DTG administered during concurrent RIF treatment and assessing safety and tolerance in HIV-TB co-infected children weighing 20 to 35 kg.

DTG will be administered as a twice-daily dose 50mg tablet formulation both before starting and after completion of the standard six-month RIF-based anti-TB treatment. The NRTI background and anti-TB drugs will be prescribed following the national weight band dosing guidelines.

Those initially diagnosed with TB are likely to be sicker, and the recommendation is to start anti-TB treatment first and follow with ART two weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Children <18 years with confirmed HIV-1 infection weighing 20-35kg ART-naive or experienced, with plans to use DTG for HIV treatment
* Diagnosis of TB disease with clinician initiating rifampicin-containing first-line therapy
* Parents/legal guardians/caregivers and children give informed written consent (or assent, where applicable) to be in the study
* Girls who have reached menses must have a negative pregnancy test at screening and be willing to adhere to two effective methods of contraception (barrier and a non-barrier form of contraception during the study, starting at least 14 days prior to enrolment) if sexually active. The parents/caregivers will be counselled together with the child if the child tests positive in order to reduce any social harm which may arise.

Exclusion Criteria:

* History or presence of known allergy or contraindications to DTG
* Alanine aminotransferase (ALT) ≥5 times the upper limit of normal (ULN), OR ALT ≥3xULN and bilirubin ≥2xULN
* Severe hepatic impairment or unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice), known biliary abnormalities (except for Gilbert's syndrome or asymptomatic gallstones)
* Pregnancy or breastfeeding
* A concurrent illness that could influence drug PK, i.e. severe diarrhoea, vomiting, renal or liver disease
* Treatment with concomitant medications known to have interactions with DTG
* Participants that are eligible for the study but refuse to give consent and/or assent

Ages: 23 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (Ctrough) of DTG 50mg twice daily | 48 weeks
  Description of the pharmacokinetics (Ctrough, Cmax and AUC0-24h) of DTG 50mg twice daily in children (20-35kg) who are taking rifampicin-based regimen for the treatment of tuberculosis.
Pharmacokinetics (Cmax) of DTG 50mg twice daily | 48 weeks
  Description of the pharmacokinetics (Cmax) of DTG 50mg twice daily in children (20-35kg) who are taking rifampicin-based regimen for the treatment of tuberculosis.
Pharmacokinetics (AUC0-24h) of DTG 50mg twice daily | 48 weeks
  Description of the pharmacokinetics (AUC0-24h) of DTG 50mg twice daily in children (20-35kg) who are taking rifampicin-based regimen for the treatment of tuberculosis.

SECONDARY OUTCOMES:
To develop an integrated model which will be used to estimate the primary PK parameters of DTG | 48 weeks
  Nonlinear mixed-effects models (NLMEM) will be used to describe the PK of DTG in an integrated model which will be used to estimate the primary PK parameters of DTG. The effect of concomitant TB treatment, as well as other covariates on these parameters, will be evaluated in the model.
Adverse events | 48 weeks
  Subjects will be monitored clinically and biologically for safety. Biological monitoring will focus on liver function. Adverse Events and Serious Adverse Events will be graded following DAIDS grading tables
Virological suppression | 48 weeks
  Antiretroviral efficacy is based on HIV viral suppression. The cut-off value related to virological failure is defined as a viral load superior to 400 copies per mL, confirmed within a month. Viral load will be assessed as per the SOE
Enzyme polymorphisms | 48 weeks
  Enzyme polymorphism analysis will be conducted at a later stage from stored samples to determine the importance of polymorphisms in genes regulating anti-TB drug and antiretroviral concentrations and effects in the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Moherndran Archary, MBChB, PhD, Principal Investigator — University of KwaZulu
Locations (1):
- King Edward VIII Hospital, Durban, KwaZulu-Natal, South Africa

REFERENCES:
- [Derived] Naidoo A, Waalewijn H, Naidoo K, Letsoalo M, Cromhout G, Sewnarain L, Mosia NR, Osuala EC, Wiesner L, Wasmann RE, Denti P, Dooley KE, Archary M; ORCHID study team. Pharmacokinetics and safety of dolutegravir in children receiving rifampicin tuberculosis treatment in South Africa (ORCHID): a prospective cohort study. Lancet HIV. 2025 Apr;12(4):e273-e282. doi: 10.1016/S2352-3018(24)00312-6. Epub 2025 Feb 26. PMID 40023169